CLINICAL TRIAL: NCT01759550
Title: Prospective Case-Series of LigaSure Advance Pistol Grip and LigaSure Blunt Tip in Gastric Procedures
Brief Title: Prospective Case-Series of Ligasure Advance Pistol Grip and LigaSure Blunt Tip
Status: Terminated | Type: Observational
Why Stopped: The Sponsor terminated the study.
Sponsor: Duke University (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00030546
Record Dates: First submitted 2012-12-31; First posted 2013-01-03 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2015-06

CONDITIONS: Morbid Obesity
Keywords: Gastric Procedures; Force Triad; LigaSure Advance Pistol Grip; LigaSure Blunt Tip
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- LigaSure Device: In this prospective observational study, 60 patients scheduled to undergo a Roux-en-Y or gastric reduction procedure (sleeve gastrectomy or plication) will have hemostasis controlled with LigaSure Advance ™ Pistol Grip or LigaSure™ Blunt Tip, respectively. Both devices are regularly used at Duke in the Bariatric Surgery division. The surgeon will select which device is used. There will be no randomization. The device decision tree will be based upon the procedure. Cases that require enterotomy will utilize the AdvanceTM pistol grip. Cases which don't need enterotomy will utilize the 5 Blunt Tip. The LigaSure AdvanceTM pistol grip and LigaSureTM Blunt Tip are used exclusively with the Force TriadTM Energy platform. There is no simultaneous use.

SUMMARY:
The study is primarily to evaluate the safety and efficacy of the LigaSure Advance™ Pistol Grip and LigaSure™ Blunt Tip using the Force Triad™ Energy Platform during Roux-en-Y and gastric reduction procedures (sleeve gastrectomy or placation), respectively. Also, Economic value of using LigaSure in gastric surgeries will be appraised.

In this prospective case series, 60 patients previously scheduled to undergo a Roux-en-Y or gastric reduction procedure (sleeve gastrectomy or placation) will have hemostasis controlled with LigaSure Advance ™ Pistol Grip or LigaSure™ Blunt Tip, respectively. All subjects undergoing Roux-en-Y or gastric reduction procedures (sleeve gastrectomy or placation) procedure at Durham Regional Hospital will be recruited.

Data Analysis will be performed using the data collected in the software program titled MetaBar at Duke University Medical Center. Categorical variables will be summarized as proportions for each category; continuous measures will be summarized by mean and standard deviation or median and range as appropriated for the data distribution. Procedure-related risks are those typically associated with gastric procedures and general anesthesia including intra-operative bleeding, infection, and injury to surrounding organs and structures. Device related risks include those normally associated with the use of electrosurgery including intra-operative bleeding, unintended tissue burns, electrical shock, and electrical stimulation of muscles and nerves.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients who will undergo a Roux-en-Y or gastric reduction procedures (sleeve gastrectomy or placation)
* Patients with a BMI between 40-60

Exclusion Criteria:

* Patients under 18 years of age
* Patients participating in other competing research protocol(s)
* Patients for whom electrosurgery is contraindicated
* Patients unable to tolerate general anesthesia
* Patients who are pregnant
* Patients unwilling or unable to provide informed consent
* Patients who have undergone significant upper GI surgery leading to adhesion formation, as determined by the Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include 60 patients previously scheduled to undergo a Roux-en-Y or gastric reduction precodures (sleeve gastrectomy or placation) using the LigaSure Advance Pistol Grip or LigaSure Blunt Tip, repectively. The pricipal investigator will be responsible for patient selection.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2011-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Safety and Efficacy of the LigaSure Advance Pistol Grip and LigaSure Blunt Tip using the Force Triad Energy Platform during Roux-en-Y and gastric reduction procedures. | 1 month
  Primary study variables include patient demographic information (age, pre- and post-operative BMI, gender, and presence of obesity associated co-morbid disease conditions such as hypertension, diabetes, sleep apnea, obesity hypoventilation, heart failure, prior blood clots, etc.), procedure time, American Society of Anesthesiologists (ASA) score, operative blood loss,length of hospital stay, and any complications noted up to one month post-operative.

SECONDARY OUTCOMES:
Economic value of using LigaSure in gastric surgeries | 1 month
  These variables include the costs of the instrument, duration and costs of anesthesia, postoperative analgesic use, and hospital day rate costs to study the economic impact of different hemostatic devices and observe trends towards cost differences. Outcomes such as perceived ergonomics, multi-functionality, and access to organs will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Portenier, MD, Principal Investigator — DUMC
Locations (1):
- Duke Center for Metabolic and Weightloss Surgery, Durham, North Carolina, United States